CLINICAL TRIAL: NCT03587948
Title: Shanghai Children and Adolescent Diabetes Eye Study
Acronym: SCADE
Status: Recruiting | Type: Observational
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018004
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus; Eye Diseases
MeSH Terms: conditions — Diabetes Mellitus; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Children and adolescents with diabetes mellitus
  Interventions: Diagnostic Test: Diabetes mellitus
- Control group: Children and adolescents without diabetes mellitus

INTERVENTIONS:
Diagnostic Test: Diabetes mellitus — Children and adolescents who is diagnosed with diabetes will be involved in case-group, and others will be involved in control-group.
  Groups: Case group

SUMMARY:
To compare the prevalence of eye disease between children and adolescents with diabetes mellitus and healthy people, and to analyze the related factors of eye diseases in diabetic patients.

DETAILED DESCRIPTION:
A cohort study. From January 2018 to 2028, 300 cases of diabetic children in Children's Hospital of Fudan University in Shanghai will be selected as case group, and 300 healthy children without diabetes will be selected as the control group.

The purpose of the study is to guide and regulate eye health screening of children and adolescents with diabetes in Children's Hospital of Fudan University in Shanghai, build up the ranks with the general practitioner as the backbone combined, and provide comprehensive, continuous, and dynamic information service to diabetic eye disease health management. We expect to reduce the prevalence rate of diabetic eye disease, blindness and visual impairment of DR, and improve diabetics consciousness of eye health maintenance, thus upgrading the level of eye disease prevention and treatment in Shanghai.

ELIGIBILITY:
Inclusion Criteria:

* (1) provision of a written informed consent by a guardian;
* (2) age over 5 years and less than 18 years;
* (3) diagnosis of type 1 or type 2 diabetes based on the WHO diagnostic criteria for cases.

Exclusion Criteria:

* (1) eyelid diseases - eyelid entropion, eyelid ectropion, eyelid, ptosis, and palpebral dyskinesia;
* (2) conjunctival diseases - pterygium and conjunctivitis;
* (3) history of ocular surface chemical injury or use of eye drops with moisturizing artificial tears;
* (4) history of eye surgery within 6 months or history of retinal laser photocoagulation;
* (5) systemic diseases - Sjogren syndrome, Parkinson's disease, rheumatoid arthritis, Grave 's disease, systemic lupus erythematosus, and others.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From January 2018 to 2028, children who are diagnosed with diabetes at the Children's Hospital of Fudan University in Shanghai, will be recruited as cases of diabetes. We will also recruit children without diabetes, who will be matched for age and gender, from this hospital as controls.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Diabetic eye diseases | January 1, 2028
  Prevalence of eye diseases due to diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, MD,PhD, Study Chair — Shanghai Eye Disease Prevention and Treatment Center
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No